CLINICAL TRIAL: NCT05747235
Title: The Role of Computed Tomography in the Phenotyping of COPD Patients
Status: Completed | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Islam Galal Sayed, Professor, Aswan University
Other Study IDs: CT in COPD phenotyping
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: CT chest — All patients will undergo MSCT chest at both inspiratory and expiratory phases in supine position without any contrast media.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common, preventable, and treatable disease that is characterized by respiratory symptoms and airflow limitation that is due to airway and/or alveolar abnormalities usually caused by significant exposure to noxious particles or gases. the CT was used for classification of COPD patients into different phenotypes: phenotype A that has minimal emphysema with or without airway disease, phenotype E that has emphysema without airway disease, and finally phenotype M as a mixed form. The investigators aimed to to identify the phenotypes of COPD using radiologic data obtained by computed tomography. Moreover, this study will be designed to answer the questions about possible correlation between pulmonary function parameters and CT.

ELIGIBILITY:
Inclusion Criteria:

* All stable COPD patients that lastly confirmed to have the disease based on spirometry and past clinical history according to GOLD (2022).
* Age above 18 years.

Exclusion Criteria:

* COPD patients associated with other chest diseases as collapse
* COPD patients associated with consolidation
* COPD patients unable to perform spirometry

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: • All stable COPD patients that lastly confirmed to have the disease based on spirometry and past clinical history according to GOLD (2022).and able to perform MSCT
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Identifying the different phenotypes of COPD using HRCT | one month
  Identifying the different phenotypes of COPD using HRCT. moreover, to identify whether there is a possible correlation between CT phenotypes and FEV1, FVC or FEV1/FVC.

CONTACTS AND LOCATIONS:
Locations (1):
- Islam Galal Sayed, Asyut, Egypt

REFERENCES:
- [Background] Fan L, Xia Y, Guan Y, Zhang TF, Liu SY. Characteristic features of pulmonary function test, CT volume analysis and MR perfusion imaging in COPD patients with different HRCT phenotypes. Clin Respir J. 2014 Jan;8(1):45-54. doi: 10.1111/crj.12033. Epub 2013 Jul 31. PMID 23711228